CLINICAL TRIAL: NCT03636685
Title: A Phase I/II Study of Anlotinib Combined With Platinum-based Chemotherapy as the First-line Treatment of Patients With Locally Advanced or Advanced Non-Small Cell Lung Cancer
Brief Title: Study of Anlotinib Plus Chemotherapy as the First-line Treatment in Patients With Advanced NSCLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shi Yuankai, Vice President of Cancer Hospital Chinese Academy of Medical Sciences, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NCC201807006
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: NSCLC; Adenocarcinoma; Squamous Cell Carcinoma
Keywords: Anlotinib; NSCLC; platinum-based chemotherapy
MeSH Terms: conditions — Adenocarcinoma; Carcinoma, Squamous Cell | interventions — Pemetrexed; Carboplatin; Clinical Trials, Phase I as Topic; Paclitaxel; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-squamous cell lung cancer (Experimental): Anlotinib combined with pemetrexed and carboplatin, phase I
  Anlotinib combined with pemetrexed and carboplatin, phase II
  Interventions: Drug: Anlotinib combined with pemetrexed and carboplatin, phase I; Drug: Anlotinib combined with pemetrexed and carboplatin, phase II
- Squamous cell lung cancer (Experimental): Anlotinib combined with paclitaxel and carboplatin, phase I
  Anlotinib combined with paclitaxel and carboplatin, phase II
  Interventions: Drug: Anlotinib combined with paclitaxel and carboplatin, phase I; Drug: Anlotinib combined with paclitaxel and carboplatin, phase II

INTERVENTIONS:
Drug: Anlotinib combined with pemetrexed and carboplatin, phase I — Non-squamous cell lung cancer, Anlotinib Plus PC
  This study will include a sequential evaluation of 3 subjects per dose group. low-dose groups: Anlotinib 8mg per day plus pemetrexed and carboplatin. middle-dose groups: Anlotinib 10mg per day plus pemetrexed and carboplatin. high-dose groups: Anlotinib 12mg per day plus pemetrexed and carboplatin to determine the appropriate dose of anlotinib in combination with paclitaxel and carboplatin
  Other Names: APC I
  Arms: Non-squamous cell lung cancer
Drug: Anlotinib combined with paclitaxel and carboplatin, phase I — Squamous cell lung cancer, Anlotinib plus TC
  This study will include a sequential evaluation of 3 subjects per dose group. low-dose groups: Anlotinib 8mg per day plus paclitaxel and carboplatin. middle-dose groups: Anlotinib 10mg per day plus paclitaxel and carboplatin. high-dose groups: Anlotinib 12mg per day plus paclitaxel and carboplatin to determine the appropriate dose of anlotinib in combination with paclitaxel and carboplatin
  Other Names: ATC I
  Arms: Squamous cell lung cancer
Drug: Anlotinib combined with pemetrexed and carboplatin, phase II — Anlotinib: established dose QD PO d1-14, pemetrexed,carboplatin, 21 days per cycle after 4-6 cycles, Anlotinib p.o, qd and it should be continued until disease progress or toxicity cannot be tolerated or patients withdraw consent
  Other Names: APCII
  Arms: Non-squamous cell lung cancer
Drug: Anlotinib combined with paclitaxel and carboplatin, phase II — Anlotinib :established dose QD PO d1-14, paclitaxel,carboplatin, 21 days per cycle
  after 4-6 cycles, Anlotinib p.o, qd and it should be continued until disease progress or toxicity cannot be tolerated or patients withdraw consent
  Other Names: ATCII
  Arms: Squamous cell lung cancer

SUMMARY:
Non-small cell lung cancer has the highest morbidity and mortality in China，and platinum-based chemotherapy is the standard first-line treatment for the wild-type NSCLC,however the overall survival still less than one year.Anlotinib is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR2、VEGFR3、PDGFRβ and c-Kit, which has strong effect of anti-angiogenesis.This study is aim to evaluate the efficacy and safety of the combination regimen of anlotinib plus platinum-based chemotherapy as first-line treatment for NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age：18~70 years;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 -2
* Subjects with histologically or cytologically confirmed locally advanced or advanced NSCLC
* EGFR\ALK\ROS1 wildtype or unknown,or patients with EGFR\ALK\ROS1 mutations but refuse to receive corresponding inhibitors' treatment
* No indications for radiation therapy
* Previously chemotherapy naive or postoperative adjuvant chemotherapy ended more than 1 year
* Subjects with at least one measurable lesion as defined by RECIST (version 1.1),which is confirmed by computed tomography (CT) scan or MRI

Exclusion Criteria:

* Small Cell Lung Cancer
* central lung squamous carcinoma along with cavum, or non-small cell lung cancer along with hemoptysis (>50ml/day)
* Within 30 days before enrollment, the patient had used any chemotherapy drugs in the previous treatment regimen or clinical study; Or, within 14 days before the first administration of the study therapy, the patient has used any targeted anticancer drugs in the previous treatment regimen or clinical study; Or stop other experimental drugs or cancer drugs for less than five half-life of the drug
* Previous use of anti-angiogenic drugs (such as anlotinib, apatinib, bevacizumab, endostar, etc.)
* have got non remissive toxic reactions derived from previous therapies, which is over level 1 in CTC AE (4.0), alopecia NOT included
* Spinal cord compression or symptomatic and untreated brain metastases (asymptomatic, stable, no need for steroid treatment for 4 weeks before study start)
* with kinds of factors which affect oral medicine (e.g. failing to swallow, gastrointestinal tract getting resected, chronic diarrhea and ileus)
* Previous histories include: interstitial pneumonia, drug-induced interstitial pneumonia, radiation pneumonia requiring steroid treatment, and clinically proven active interstitial pneumonia
* get arterial/venous thrombosis within 6 months, such as cerebrovascular accidents (including temporary ischemic stoke), prevenous thrombosis, and pulmonary embolism
* Have suffered from hemorrhagic disease or coagulation dysfunction
* diagnosed with disease which will severely endanger the security of patients or influence the completion of this research

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2019-08-14 (Estimated); Study Completion 2020-08-14 (Estimated)

PRIMARY OUTCOMES:
Progress free survival (PFS) | From date of enrollment until the date of first documented progression or date of death from any cause,whichever came first.up to 12 months
  progression free survival

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | each 21 days up to the toxicity or PD (up to 24 months)
  Objective Response Rate
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Disease Control Rate
Overall Survival (OS) | From enrollment until death (up to 36 months)
  Overall survival
Number of Participants with Adverse Events as a Measure of Safety and Tolerability (Safety) | Time Frame: each 21 days up to the toxicity or PD (up to 36 months)
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Han B, Li K, Zhao Y, Li B, Cheng Y, Zhou J, Lu Y, Shi Y, Wang Z, Jiang L, Luo Y, Zhang Y, Huang C, Li Q, Wu G. Anlotinib as a third-line therapy in patients with refractory advanced non-small-cell lung cancer: a multicentre, randomised phase II trial (ALTER0302). Br J Cancer. 2018 Mar 6;118(5):654-661. doi: 10.1038/bjc.2017.478. Epub 2018 Feb 13. PMID 29438373